CLINICAL TRIAL: NCT03744299
Title: The Interest of Cancer Patients and Caregivers in Acupuncture: a Survey
Acronym: ACTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Principal investigator, General Hospital Groeninge
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AZGS2018093
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2018-11

CONDITIONS: Cancer
Keywords: acupuncture; surveys and questionnaires; patient; caregiver
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Patients and caregivers are asked to complete a questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients and caregivers are asked to complete a questionnaire

SUMMARY:
Cancer and cancer treatments are accompanied by several possible side effects, such as nausea, hot flashes, fatigue, drowsiness, etc. Complementary and integrative therapies, such as acupuncture, could be used to manage these symptoms. The aim of this study for our research team is to have an idea of the interest of cancer patients and caregivers in acupuncture. This is a prospective, interventional study. Cancer patients and caregivers will be approached at the day care clinic by a health care worker to participate in this study. They will be asked to complete a questionnaire about their interest in acupuncture and their motivation, what symptoms they would need it for, where they would like this acupuncture to take place, whether they are willing to pay for it, and whether they would be interested in an information session about acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Dutch speaking patients and caregivers
* Patients and caregivers presenting at the outpatient clinic, including the day-care clinic and follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Response rate | At study inclusion

SECONDARY OUTCOMES:
Interest in acupuncture assessed by questionnaire | At study inclusion
Side effects participants would like to receive acupuncture for assessed by questionnaire | At study inclusion
Place where an acupuncture treatment should take place assessed by questionnaire | At study inclusion
Willingness to pay for an acupuncture treatment assessed by questionnaire | At study inclusion
Interest in an information session about acupuncture assessed by questionnaire | At study inclusion
Patient or caregiver characteristics (sex, age, diagnosis) collected by questionnaire | At study inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Philip Debruyne, MD, PhD, MSc, FRCP, Principal Investigator — General Hospital Groeninge
Locations (1):
- General Hospital Groeninge, Cancer Center, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No